CLINICAL TRIAL: NCT06716125
Title: Lifestyle Changes in Obese Males With Sexual Dysfunction and Tinnitus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, Department of Physical Therapy for Cardiovascular/Respiratory Disorder and Geriatrics, Faculty of Physical Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00014233-16
Record Dates: First submitted 2024-11-28; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Obesity; Tinnitus, Subjective; Erectile Dysfunction
MeSH Terms: conditions — Obesity; Tinnitus; Erectile Dysfunction | interventions — Caloric Restriction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group I (Experimental): This group (n =20 for the group) will administer low calorie diet for 12 weeks plus additionally administering supervised walking training aerobic training for 45 minutes 3 times per week for 12 weeks.
  Interventions: Behavioral: aerobic treadmill walking plus low calorie diet
- Group II (Active Comparator): this group (n =20 for the group) will administer low calorie diet for 12 weeks
  Interventions: Behavioral: low calorie diet

INTERVENTIONS:
Behavioral: aerobic treadmill walking plus low calorie diet — this group (n =20 for the group) will administer low calorie diet for 12 weeks plus additionally administering supervised walking treadmill aerobic training for 45 minutes 3 times per week for 12 weeks).
  Arms: group I
Behavioral: low calorie diet — this group (n =20 for the group) will administer low calorie diet for 12 weeks
  Arms: Group II

SUMMARY:
obese male usually complain subjective tinnitus that may affect their sexual function.

DETAILED DESCRIPTION:
this study will enroll forty obese males with subjective tinnitus (bilateral complaint) and sexual dysfunction (erectile dysfunction) who will be divided to group I and group II with an equal number of males within each group (n =20 for the group). all male in both groups will administer low calorie diet for 12 weeks but Group I will additionally administer supervised walking training aerobic training for 45 minutes 3 times per week for 12 weeks).

ELIGIBILITY:
Inclusion Criteria:

* obese person
* body mass index less than 40 kg/m2 and more than 30 kg/m2
* males with subjective tinnitus (bilateral presentation from at least 24 weeks).
* males with sexual dysfunction (erectile dysfunction from at least 24 weeks)

Exclusion Criteria:

* cardiac diseased males
* respiratory diseased males
* hepatic, musculoskeletal, and hepatic diseased males
* diabetic males

Ages: 35 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — based on self-representation of gender identity.
Enrollment: 40 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2025-04-06 (Estimated); Study Completion 2025-04-06 (Estimated)

PRIMARY OUTCOMES:
international index of erectile function | it will be assessed after 12 weeks
  Arabic form that contain five question will be used

SECONDARY OUTCOMES:
body mass index | it will be assessed after 12 weeks
  it will be assessed at empty stomach and bladder
waist circumference | it will be assessed after 12 weeks
  it will be assessed at level of umbilicus
visual analogue scale of severity of tinnitus | it will be assessed after 12 weeks
  it will be 10-cm line that will be used to assess tinnitus severity
visual analogue scale of discomfort induced by tinnitus | it will be assessed after 12 weeks
  it will be 10-cm line that will be used to assess discomfort induced by tinnitus
tinnitus handicap inventory | it will be assessed after 12 weeks
  it is a questionnaire that will assess quality of life impacted by tinnitus
triglycerides | it will be measured after 12 weeks
  it will be measured in plasma
high density lipoprotein | it will be measured after 12 weeks
  it will be measured in plasma
atherogenic index | it will be measured after 12 weeks
  it will be assessed as and indicator of atherosclerotic status

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- faculty of physical therapy Cairo university, Dokki, Giza Governorate, Egypt